CLINICAL TRIAL: NCT05677906
Title: Rural Libraries Promoting Walking and Walkability in Their Rural Communities
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Texas A&M University (Other); University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00024665
Record Dates: First submitted 2022-12-07; First posted 2023-01-10 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Physical Activity
Keywords: rural populations; physical activity promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking only (Step It Up!) (Active Comparator): A group-based, weekly walking program (Step It Up) where participants walk for up to 45 minutes.
  Interventions: Other: Walking only (Step It Up!)
- Combined (Step It Up! plus Change Club) (Experimental): A group-based, weekly walking program (Step It Up) where participants walk for up to 45 minutes. Participants also spend 30 minutes each week in a civic engagement program (the Change Club) improving walkability in the community
  Interventions: Other: Walking only (Step It Up!); Other: Combined (Step It Up! plus Civic Engagement)

INTERVENTIONS:
Other: Walking only (Step It Up!) — Participants will meet weekly for 60 minutes and walk together as a group. Participants will progressively build up to walking for 45 minutes at a brisk pace. Walks will start with a check-in and end with stretching as a group.
Other: Combined (Step It Up! plus Civic Engagement) — Participants in the combined groups will meet weekly for 90 minutes with group members. They will participate in a group walk for 60 minutes followed by 30 minutes of civic engagement aimed at improving walkability in the community
  Arms: Combined (Step It Up! plus Change Club)

SUMMARY:
The investigators will randomize 20 rural libraries to implement either a group-based walking (standard approach) or a group-based walking combined with a civic engagement program (combined approach). Each rural library will enroll between 15-20 participants. The investigators will compare the change in physical activity between participants in each group.

DETAILED DESCRIPTION:
The goals of this study are:

1. Increase the capacity of rural libraries to deliver evidence-based health promotion programs
2. Compare the effects of a group-based walking program with a combined group-based plus civic engagement program on physical activity, cardiovascular fitness and collective efficacy among rural residents.
3. Evaluate program implementation

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Inactive (defined as engaging in physical activity <3 days per week)
* Ability to walk for at least 20 minutes
* Living within the rural community served by the local library
* Ability to travel to the local library/location of walking group.

Exclusion criteria:

* Participation/intention to participate in other lifestyle modification pro-gram(s)
* Cognitive impairment
* Inability to communicate due to severe uncorrected hearing loss or speech disorder or severe visual impairment (if precludes completion of assessments and/or intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Change from baseline physical activity at 6 months, 12 months, and 24 months.
  Participants will be asked to wear an accelerometer for >10 hours/day for seven days at the wrist to measure physical activity. An accelerometer is a small device worn at the wrist that records acceleration, the change in velocity of a participant over time.
Cardio respiratory fitness | Change from baseline cardio respiratory fitness at 6 months, 12 months, and 24 months.
  Participants will be asked to complete a six-minute walk test to measure cardiorespiratory fitness. The distance walked in 6 minutes will be recorded.
Collective Efficacy | Change from baseline collective efficacy at 6 months, 12 months, and 24 months
  Participants will be asked to complete a survey regarding collective-efficacy, the Collective Efficacy Scale (Sampson and colleagues, 1997), which measures how well communities work together to make things happen.

SECONDARY OUTCOMES:
Height | Baseline
  Researchers will measure the height of participants in inches.
Hip circumference | Change from baseline hip circumference at 6 months, 12 months, and 24 months.
  Researchers will measure the hip circumference of participants in inches.
Resting heart rate | Change from baseline resting heart rate at 6 months, 12 months, and 24 months.
  Researchers will measure resting heart rate of participants by using heart rate monitor.
Weight | Change from baseline weight at 6 months, 12 months, and 24 months.
  Researchers will measure the weight of participants in pounds.
Blood pressure | Change from baseline blood pressure at 6 months, 12 months, and 24 months.
  Researchers will measure the both diastolic and systolic blood pressure of participants using a sphygmomanometer.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia K Perry, PhD, Principal Investigator — Oregon Health & Science University School of Nursing
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will involve the collection of qualitative and quantitative data. The investigators will not share the qualitative data due to the potential to compromise participant identity and related ethical concerns. Quantitative data from the participants will include demographic, anthropometric, physiologic, and behavioral data. Identifiers will be removed from the final datasets prior to release for sharing. However, given the small populations of the targeted communities, data will only be made available through a data sharing agreement to prevent the possibility of identity disclosure. This agreement will ensure that the data are used for research purposes only, that it will be kept secure, and that it will be destroyed or returned following analysis completion.
Time Frame: Data will become available once all manuscripts have been published.
Access Criteria: Data will be made available through a data sharing agreement.

REFERENCES:
- [Background] Lenstra N. The role of public librarians in supporting physical activity: challenging the "Jacks of All Trades but Masters of None" librarian syndrome. Advances in Library Administration and Organization. 2018;39:185-205.
- [Background] Perry CK, Campbell LP, Currier J, Farris PE, Wenzel ES, Medysky ME, Zell A, McDonell M, Shannon J, Winters-Stone K. An Evidence-Based Walking Program in Oregon Communities: Step It Up! Survivors. Prev Chronic Dis. 2020 Dec 10;17:E156. doi: 10.5888/pcd17.200231. PMID 33301392
- [Background] Seguin RA, Sriram U, Connor LM, Silver AE, Niu B, Bartholomew AN. A Civic Engagement Approach to Encourage Healthy Eating and Active Living in Rural Towns: The HEART Club Pilot Project. Am J Health Promot. 2018 Sep;32(7):1591-1601. doi: 10.1177/0890117117748122. Epub 2018 Feb 1. PMID 29390863
- [Derived] Perry CK, Seguin-Fowler R, Maddock JE, Lenstra N, Dieckmann NF, Currier J, Andreyeva E, Winkle J, Trost SG. Rural libraries implementing walking groups or walking groups plus civic engagement for walkability in rural communities: a comparative effectiveness trial study protocol. BMC Public Health. 2023 Oct 2;23(1):1895. doi: 10.1186/s12889-023-16788-0. PMID 37784086